CLINICAL TRIAL: NCT02746315
Title: A Randomised, Double-blind, Single-centre, Placebo-controlled, Dose Escalation, Multiple s.c. DoseStudy to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HS-20004 in Healthy Chinese Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple s.c Doses HS-20004 in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-20004-Ib
Record Dates: First submitted 2016-04-11; First posted 2016-04-21 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Experimental 1 (Experimental): Once daily subcutaneous dose for 7 Days of HS-20004 0.02 mg or Matched Placebo.
  Interventions: Drug: HS-20004; Drug: Placebo
- Experimental 2 (Experimental): Once daily subcutaneous dose for 7 Days of HS-20004 0.04 mg or Matched Placebo.
  Interventions: Drug: HS-20004; Drug: Placebo
- Experimental 3 (Experimental): Once daily subcutaneous dose for 7 Days of HS-20004 0.06 mg or Matched Placebo.
  Interventions: Drug: HS-20004; Drug: Placebo
- Experimental 4 (Experimental): Once daily subcutaneous dose for 7 Days of HS-20004 0.08 mg or Matched Placebo.
  Interventions: Drug: HS-20004; Drug: Placebo

INTERVENTIONS:
Drug: HS-20004
Drug: Placebo

SUMMARY:
This trial is conducted in China. The aim of this trial is to assess the safety and tolerability for Multiple s.c injection of HS-20004 in healthy Chinese subjects

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 19 and 28 kg/m^2, inclusive, and a total body weight of at least 50 kg;

Exclusion Criteria:

* Clinically relevant abnormalities of physical examination, laboratory values, vital signs or ECG findings at the screening, as judged by the Investigator;
* Have any other medical abnormality (such as cardiovascular, hepatic, renal, gastrointestinal, immunologic, hematological, hormonal, metabolic, neoplasmatic or mental disease), which in the opinion of the investigator, might affect the absorption, distribution, metabolism, and excretion of the study drug, or prevent the patient from following and completing the protocol;
* Family history of diabetes, thyroid cancer, submandibular gland cancer, or history of pancreatitis, cholelithiasis, drug allergy, serious unconscious hypoglycemia or positive of anxious chronic viral hepatitis B, HIV antibody;
* History of drug or alcohol abuse within 6 months before randomization;
* Use of GLP-1 analogues, DPP-IV enzyme inhibitors, as well as other hypoglycemic drugs within 3 months before randomization;
* Use of any prescription drugs and Chinese herbal medicines within 4 weeks before randomization;
* Use of non prescription drugs and food supplements (vitamins, etc.) within 2 weeks before randomization;
* Participated any drug clinical trials within 3 months, or participated 3 or more than 3 drug clinical trials within 1 year, or had blood donation/loss >400mL within 3 months before randomization;
* Female subject of childbearing potential who does not use an acceptable method of birth control, is pregnant or planning a pregnancy, or breastfeeding, or male subject who does not use an acceptable method of birth control, within six months before randomization;
* Subject who cannot refrain from smoking, eating and/or drinking containing xanthine/caffeine, or strenuous exercise, or others that affect drug absorption, distribution, metabolism and excretion within 2 days before the study drug administration; Subject who is unsuitable for inclusion in the study in the opinion of the investigator;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10; Primary Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | Day 0 and up to 3 days after last treatment (Day 10)

SECONDARY OUTCOMES:
Area under the plasma HS-20004 concentration curve after the last s.c injection | Time 0 to 72 hours after the last dose
Peak plasma concentration (Cmax) after the last dose | Time 0 to 72 hours after the last treatment
Terminal elimination half-life (t½) for HS-20004 after the last dose | Time 0 to 72 hours after the last treatment
Change in 24-hour profiles of plasma glucose and serum insulin from baseline | From time 0 to 24 hours after the first and last treatment

IPD SHARING:
Plan to Share IPD: No